CLINICAL TRIAL: NCT02598661
Title: A Study to Evaluate Imetelstat (GRN163L) in Transfusion-Dependent Subjects With IPSS Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS) That is Relapsed/Refractory to Erythropoiesis-Stimulating Agent (ESA) Treatment
Brief Title: Study to Evaluate Imetelstat (GRN163L) in Participants With International Prognostic Scoring System (IPSS) Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107947; 63935937MDS3001 (Other: Geron); EU CTIS number (Other: 2024-511348-25-00); 2015-002874-19 (EudraCT Number)
Record Dates: First submitted 2015-10-27; First posted 2015-11-06 (Estimated); Results first posted 2025-02-14 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Imetelstat Sodium; GRN163L; Relapsed/refractory to ESAs; Transfusion dependent; IMerge
MeSH Terms: conditions — Myelodysplastic Syndromes; Recurrence | interventions — imetelstat; GRN163L peptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 2: Imetelstat Sodium (Experimental): Imetelstat sodium administered intravenously (IV), at a starting dose of 7.5 milligrams per kilogram (mg/kg), every 4 weeks (on a 28-day cycle) until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first. Dose escalation to 9.4 mg/kg was allowed before Protocol Amendment 2.
  Interventions: Drug: Imetelstat Sodium
- Phase 3: Imetelstat Sodium (Experimental): Imetelstat sodium administered IV, at a starting dose of 7.5 mg/kg, every 4 weeks (on a 28-day cycle) until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first.
  Interventions: Drug: Imetelstat Sodium
- Phase 3: Placebo (Placebo Comparator): Imetelstat sodium-matching placebo administered IV, every 4 weeks (on a 28-day cycle), until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first.
  Interventions: Drug: Placebo
- QTc Substudy: Imetelstat Sodium (Experimental): Imetelstat sodium administered IV, at a starting dose of 7.5 mg/kg, every 4 weeks (on a 28-day cycle) until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first.
  Interventions: Drug: Imetelstat Sodium
- QTc Substudy: Placebo (Placebo Comparator): Imetelstat sodium-matching placebo administered IV, every 4 weeks (on a 28-day cycle), until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first. If after a minimum of 2 treatment cycles a participant has no significant change to pRBC transfusion burden or evidence of clinical benefit per Investigator, after discussion with the Sponsor the participant, he/she may be permitted to start treatment with imetelstat sodium.
  Interventions: Drug: Placebo
- Extension Phase: Imetelstat Sodium (Experimental): Participants randomized to the imetelstat sodium arm in the Phase 3 and the VR QTc Substudy, based on the response will continue to receive imetelstat sodium IV, at the dose they were receiving in the Phase 3 or VR QTc Substudy, every 4 weeks (on a 28-day cycle) until death, lost to follow-up, withdrawal of consent, study termination, or up to 3 years whichever occurs first.
  Interventions: Drug: Imetelstat Sodium
- Extension Phase: Extended Follow-up (Experimental): Participants randomized to the placebo arm in the Phase 3 study will enter the Extended Follow-up part of the Extension Phase and continue in follow up until death, lost to follow-up, withdrawal of consent, study termination, or whichever occurs first up to approximately 3 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imetelstat Sodium — Imetelstat sodium IV infusion.
  Other Names: GRN163L
  Arms: Extension Phase: Imetelstat Sodium; Phase 2: Imetelstat Sodium; Phase 3: Imetelstat Sodium; QTc Substudy: Imetelstat Sodium
Drug: Placebo — Imetelstat sodium-matching placebo IV infusion.
  Arms: Extension Phase: Extended Follow-up; Phase 3: Placebo; QTc Substudy: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of imetelstat sodium in transfusion-dependent participants with low or intermediate-1 risk myelodysplastic syndrome (MDS) that is relapsed/refractory to erythropoiesis-stimulating agent (ESA) treatment in Phase 2 study and to compare the efficacy, in terms of red blood cell (RBC) transfusion independence (TI), of imetelstat sodium to placebo in transfusion-dependent participants with low or intermediate-1 risk MDS that is relapsed/refractory to ESA treatment in Phase 3 study.

A separate Ventricular Repolarization Substudy (QTc Substudy) will evaluate the effect of imetelstat sodium on ventricular repolarization.

An Extension Phase has been included to allow continued treatment for those participants who are benefitting from imetelstat sodium and to continue to evaluate the long-term safety, overall survival (OS), and disease progression, including progression to acute myeloid leukemia (AML) in transfusion-dependent participants with low or immediate-1 risk MDS that is relapsed/refractory to ESA treatment.

DETAILED DESCRIPTION:
This is a Phase 2/3, multicenter study of imetelstat sodium in which 289 participants were enrolled.

* Phase 2 is an open-label, single-arm design to assess the efficacy and safety of imetelstat sodium. A total of 57 participants were enrolled in Phase 2, including the expansion cohort.
* Phase 3 is a double-blind, randomized design to compare the efficacy of imetelstat sodium with placebo. In the Phase 3 study, 178 participants were enrolled and randomized in a 2:1 ratio to receive either imetelstat sodium or placebo, respectively.
* In a separate Ventricular Repolarization (VR) Substudy (QTc Substudy), 54 participants were enrolled and randomized 2:1 to receive either imetelstat sodium or placebo. If after a minimum of 2 treatment cycles in the VR substudy, a participant has no significant change to packed red blood cell (pRBC) transfusion burden or evidence of clinical benefit per Investigator, after discussion with the Sponsor the participant may be unblinded. If the participant was on placebo treatment, he/she may be permitted to start treatment with imetelstat sodium.

The Extension Phase was initiated at the end of the Phase 3 study (24 months after the last participant was randomized in the Phase 3) and will continue until participants who entered Phase 3 study participated in the study for up to 5 years from the first dose of imetelstat sodium (including treatment and follow-up), or 3 years of post-treatment follow-up from the last dose of study treatment, whichever occurs later, or until death, withdrawal of consent, study termination, or until a participant is lost to follow-up. Participants ongoing on imetelstat sodium and considered to be benefiting from treatment per Investigator in the Phase 3 Study or Ventricular Repolarization Substudy, have the option to continue receiving imetelstat sodium in the Extension Phase. Participants in the follow-up phase for the Phase 3 study or Ventricular Repolarization Substudy have the option to continue the follow-up in the Extension Phase.

The Phase 2, Phase 3, and VR Substudy all consist of 3 phases: a Screening phase (up to 28 days); a treatment phase; and a post-treatment follow-up phase which will continue until death, lost to follow-up, withdrawal of consent, or the End of the Study (whichever occurs first). The Extension Phase of the study will consist of an extended treatment phase and an extended follow-up phase which will continue until death, lost to follow-up, withdrawal of consent, or the End of the Study (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman greater than or equal to (≥) 18 years of age
* Diagnosis of myelodysplastic syndrome (MDS) according to World Health Organization (WHO) criteria confirmed by bone marrow aspirate and biopsy within 12 weeks prior to Cycle 1 Day 1 (C1D1) (Phase 2) or randomization (Phase 3). In Ventricular Repolarization Substudy, diagnosis of MDS or myelodysplastic/myeloproliferative neoplasm with ring sideroblasts and thrombocytosis (MDS/MPN-RS-T) according to WHO criteria confirmed by bone marrow aspirate and biopsy within 12 weeks prior to C1D1
* International Prognostic Scoring System (IPSS) low Risk or intermediate-1 risk MDS
* Red blood cell (RBC) transfusion dependent, defined as requiring at least 4 RBC units transfused over an 8-week period during the 16 weeks prior to Study Entry; pre-transfusion hemoglobin (Hb) should be less than or equal to (≤) 9.0 gram per deciliter (g/dL) to count towards the 4 units total
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2

Exclusion Criteria:

* Participant has known allergies, hypersensitivity, or intolerance to imetelstat sodium or its excipients
* Participant has received an investigational drug or used an invasive investigational medical device within 30 days prior to Study Entry or is currently enrolled in an investigational study
* Prior treatment with imetelstat sodium
* Have received corticosteroids greater than (>) 30 milligram per day (mg/day) prednisone or equivalent, or growth factor treatment within 4 weeks prior to study entry
* Has received an erythropoiesis-stimulating agent (ESA) or any chemotherapy, immunomodulatory, or immunosuppressive therapy within 4 weeks prior to study entry (8 weeks for long-acting ESAs)
* Phase 3: a) Prior treatment with a hypomethylating agent (example [eg], azacitidine, decitabine); b) Prior treatment with lenalidomide

Additional Exclusion Criteria for the Ventricular Repolarization Substudy:

* Concurrent therapy with medications known to prolong the QT interval and have been associated with Torsade de pointes arrhythmia (TdP)
* Cardiac function abnormalities on screening ECG as follows:

  * Resting heart rate outside of 50 to 100 beats per minute
  * QT interval by Fridericia's correction method (QTcF) >470 millisecond (msec) (or QTcF >490 msec in the presence of a right bundle branch block or ventricular conduction delay [QRS >119 msec]), determined by central assessment based on the average value of a triplicate set of ECGs
  * Diagnosed or suspected congenital long QT syndrome
  * Family history of sudden unexpected death from cardiac-related causes if indicative of a pathogenic mutation of cardiac ion channels
  * Family history of congenital long QT syndrome
  * History of Mobitz II second degree or third degree heart block
  * Implantable pacemaker or automatic implantable cardioverter defibrillator
  * Complete left bundle branch block
  * Chronic or persistent atrial arrhythmia including atrial fibrillation and atrial flutter
  * History or presence of clinically relevant heart rhythm disturbances including atrial, junctional, re-entry, and ventricular tachycardia
  * Unusual T-wave morphology (i.e., bifid T-wave) likely to interfere with QT measurements
* History or evidence for any of the following: severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (example, pulmonary embolism, cerebrovascular accident including transient ischemic attacks) within 12 months prior to Cycle 1 Day 1, New York Heart Association (NYHA) Class II to IV heart disease
* Presence of uncontrolled hypertension (persistent systolic blood pressure [BP] ≥160 mmHg or diastolic BP ≥100 mmHg). Participants with a history of hypertension are permitted, provided that BP is controlled to within these limits by anti-hypertensive treatment
* Any skin condition likely to interfere with electrocardiographic electrode placement or adhesion
* History of thoracic surgery likely to cause abnormality of the electrical conduction through thoracic tissues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2026-10-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tymara Berry, MD, Study Director — Geron Corporation
Locations (126):
- United States (22):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Acrc/Arizona Clinical Research, Inc., Tucson, Arizona
  - CBCC Global Research, Inc., Bakersfield, California
  - UCLA Ronald Regan Medical Center, Los Angeles, California
  - Yale-New Haven Hospital (YNHH) - Smilow Cancer Hospital, New Haven, Connecticut
  - BRCR Medical Center, Plantation, Florida
  - University of South Florida (USF) - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Franciscan Health, Indianapolis, Indiana
  - St. Agnes Healthcare, Inc, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai Program for the Protection of Human Subjects, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic Taussig Cancer, Cleveland, Ohio
  - The Ohio State Comprehensive Cancer Center, Columbus, Ohio
  - Prairie lakes Healthcare system, Inc, Watertown, South Dakota
  - Vanderbilt University Medical - Hematology-Oncology, Nashville, Tennessee
  - Texas Oncology/Methodist Charlton Cancer Center, Dallas, Texas
  - Simmons Comprehensive Cancer Center, Dallas, Texas
  - Fred Hutchinson Cancer Research Center (FHCRC), Seattle, Washington
- Belgium (8):
  - ZAS Middelheim, Antwerp, Antwerpen
  - ZAS Cadix, Antwerp, Antwerpen
  - GZA Ziekenhuizen - Campus Sint, Wilrijk, Antwerpen
  - AZ Sint-Jan Burgge-Oostende, Bruges, West-Vlaanderen
  - Az Groeninge, Kortrijk, West-Vlaanderen
  - AZ Klina, Brasschaat
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven - Campus Gasthuisberg, Leuven
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital - Hematology Research, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Brno, Brno, Brno-město
  - FN Hradec Kralove, Hradec Králové, Hradec Králové
  - FN Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (10):
  - Hopital de l'Archet, Nice, Alpes-Maritimes
  - CHU Tours, Tours, Centre-Val de Loire
  - CHU de Limoges, Hopital Dupuytren, Limoges, Haute-Vienne
  - CHU de Grenoble - Hôpital Albe, La Tronche, Isère
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CH Le Mans - HAEMATOLOGY, Le Mans, Sarthe
  - CHU de Poitiers, Poitiers, Vienne
  - Centre Hospitalier Universitai, Angers
  - CHRU de Lille - Hopital Claude Huriez - Maladies du Sang, Lille
  - CHU - HÃ´pital Saint Louis - H, Paris, Île-de-France Region
- Germany (8):
  - University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Fachärztliche Gemeinschaftspraxis mit Schwerpunkt, Dresden, Saxony
  - University Hospital Leipzig, Leipzig, Saxony
  - Studienzentrum für Hämatologie, Onkologie,Diabetologie, Endoskopie und Fußambulanz, Aschaffenburg
  - University Hospital Bonn, Bonn
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Johannes Gutenberg Universität, Mainz
- Israel (9):
  - The Edith Wolfson Medical Center, H̱olon, Central District
  - Meir Medical Center, Kfar Saba, Central District
  - Kaplan Medical Center, Rehovot, Hagalil Saint
  - Hadassah Medical Organization, Jerusalem, Jerusalem
  - Ha'Emek Medical Center, Afula, Northern District
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky, Tel Aviv
  - Carmel MC, Haifa
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
- Italy (10):
  - A.O. Ospedale Niguarda Ca' Granda, Milan, Lombardy
  - Istituto Clinico Humanitas Rozzano, IRCCS, Rozzano, Milano
  - Irccs Crob, Rionero in Vulture, Potenza
  - A.O. Universitaria Policlinico Tor Vergata, Roma, Roma
  - AOU Ospedali Riuniti Umberto I G.M. Lancisi G. Salesi, Ancona
  - AOU di Bologna Policlinico S. Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi di Firenze, Florence
  - Grande Ospedale Metropolitano 'Bianchi-Melacrino-Morelli' Reggio Calabria, Reggio Calabria
  - AO S. Andrea, Università degli Studi di Roma La Sapienza, Roma
  - Ospedale di Circolo, PO Varese, Varese
- Netherlands (4):
  - Radboud Umcn, Nijmegen, Gelderland
  - Meander Medisch Centrum, Amersfoort
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- Poland (5):
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego, Wroclaw, Lower Silesian Voivodeship
  - Wojewódzki Szpital Specjalistyczny sp.z o.o., Słupsk, Pomeranian Voivodeship
  - PRATIA Poznań, Poznan, Ul. Gryfińska 1
  - SPZOZ MSWiA z Warminsko - Mazurskim Centrum Onkologii, Olsztyn, Warmian-Masurian Voivodeship
  - Ars Medical sp. z o.o., Piła, Wielkopolskie Województwo
- Russia (7):
  - Clinics of Samarskiy GMU, Samara, Volga
  - Emergency Hospital of Dzerzhinsk, Dzerzhinsk
  - City Clinical Hospital, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Ryazan Regional Clinical Hospital, Ryazan
  - FGU-Russian Research Institut, Saint Petersburg
  - Oncologic Dispensary No.2, Sochi
- South Korea (8):
  - Pusan National University Hospital - Hematology and Oncology, Seogu, Incheon
  - Gachon University Gil Medical Center - oncology, Incheon, Incheon Gwang'Yeogsi
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei Uni, Seoul
- Spain (11):
  - H.U.Pta.del Mar, Cadiz, Cádiz
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Nuestra Señora de Valme, Seville, Sevilla
  - Hospital Universitario Doctor, Valencia, Valencia
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Clinico Univ. de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe, Valencia
- Switzerland (4):
  - University Hospital in Basel, Basel, Basel-Stadt (de)
  - Inselspital - Universitätsspital Bern, Bern, Canton of Bern
  - Kantonsspital St. Gallen - Onkologie/Hämatologie, Sankt Gallen, Canton of St. Gallen
  - Universitaetsspital Zuerich, Zurich, Canton of Zurich
- Turkey (Türkiye) (3):
  - Ankara University Medical Faculty - Hematology, Ankara, Anatolia
  - Ege Universitesi Tip Fakultesi - Hematology, Izmir, İzmir
  - Cukurova University Medical Faculty, Adana
- Ukraine (3):
  - KNP "Cherkaskyi oblasnyi onkolohichnyi dyspanser Cherkaskoi, Cherkasy, Cherkasy Oblast
  - KZ "Miska bahatoprofilna klinichna likarnia No4", hematolohi, Dnipro, Dnipropetrovsk Oblast
  - Instytut patolohii krovi ta transfusiynoi medytsyny NAMN Ukr, Lviv, Lviv Oblast
- United Kingdom (4):
  - The Leeds Teaching Hospitals NHS Trust, Leeds, Leeds
  - Nottingham City Hospital - Clinical Haematology, Nottingham, Nottinghamshire
  - Southampton University Hospital, Southampton, Southampton
  - Aberdeen Royal Infirmary, Aberdeen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim N, Pulte ED, Ehrlich LA, Ionan AC, Haupert S, Vallejo J, Green F, Zheng N, Wang Y, Liu J, Blanco JG, Dorff SE, Booth B, Choe M, Gehrke B, Bhatnagar V, Theoret M, Pazdur R, De Claro RA, Norsworthy KJ. US Food and Drug Administration Approval Summary: Imetelstat for Selected Patients With Low- to Intermediate-1 Risk Myelodysplastic Syndromes With Transfusion-Dependent Anemia. J Clin Oncol. 2025 Dec 10;43(35):3760-3768. doi: 10.1200/JCO-25-01369. Epub 2025 Oct 24. PMID 41135032
- [Derived] Platzbecker U, Santini V, Fenaux P, Sekeres MA, Savona MR, Madanat YF, Diez-Campelo M, Valcarcel D, Illmer T, Jonasova A, Belohlavkova P, Sherman LJ, Berry T, Dougherty S, Shah S, Xia Q, Sun L, Wan Y, Huang F, Ikin A, Navada S, Feller F, Komrokji RS, Zeidan AM. Imetelstat in patients with lower-risk myelodysplastic syndromes who have relapsed or are refractory to erythropoiesis-stimulating agents (IMerge): a multinational, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2024 Jan 20;403(10423):249-260. doi: 10.1016/S0140-6736(23)01724-5. Epub 2023 Dec 1. PMID 38048786
- [Derived] Steensma DP, Fenaux P, Van Eygen K, Raza A, Santini V, Germing U, Font P, Diez-Campelo M, Thepot S, Vellenga E, Patnaik MM, Jang JH, Varsos H, Bussolari J, Rose E, Sherman L, Sun L, Wan Y, Dougherty S, Huang F, Feller F, Rizo A, Platzbecker U. Imetelstat Achieves Meaningful and Durable Transfusion Independence in High Transfusion-Burden Patients With Lower-Risk Myelodysplastic Syndromes in a Phase II Study. J Clin Oncol. 2021 Jan 1;39(1):48-56. doi: 10.1200/JCO.20.01895. Epub 2020 Oct 27. PMID 33108243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in Phase 2 at 48 study sites and in the Phase 3 Study at 77 study sites. Data is reported for the Phase 2, Phase 3 and QTc substudy up to the primary completion date (PCD) of 13 October 2023. Enrolment in Extension phase started after October 2023 and analyses for the participants in extension phase is still ongoing, hence data for extension phase will be reported at study completion date in 2026.
Pre-assignment Details: 57 participants with MDS received Imetelstat Sodium in Phase 2, followed by Phase 3 where 178 participants were randomized to receive either Imetelstat Sodium or Imetelstat sodium-matching placebo. 54 participants enrolled in QTc Substudy to receive either Imetelstat Sodium or Imetelstat sodium-matching placebo.
Period: Overall Study
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo | QTc Substudy: Imetelstat Sodium | QTc Substudy: Placebo
Started | 57 | 118 | 60 | 35 | 19
Crossover to Imetelstat | 0 | 0 | 0 | 0 | 14
Target Population (The Target Population included the participants without prior hypomethylating agent (HMA) or lenalidomide use and non del(5q) in karyotype at baseline.) | 38 | 0 | 0 | 0 | 0
Completed | 15 | 57 | 29 | 33 | 17
Not Completed | 42 | 61 | 31 | 2 | 2
Not completed — Death | 27 | 34 | 14 | 1 | 0
Not completed — Lost to Follow-up | 2 | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 24 | 14 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Randomized, Never Treated | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Phase 2: All Treated Analysis Set included all participants who received at least one dose of study drug. Phase 3: Intent-to-Treat (ITT) Analysis Set included all participants randomized into the phase 3 study. The QTc Substudy Analysis Set included all participants who participated in QTc Substudy and received at least one dose of study drug.
Groups:
- Phase 2: Imetelstat Sodium: Imetelstat sodium administered IV, at a starting dose of 7.5 mg/kg, every 4 weeks (on a 28-day cycle) until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first. Dose escalation to 9.4 mg/kg was allowed before Protocol Amendment 2.
- Total: Total of all reporting groups
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo | QTc Substudy: Imetelstat Sodium | QTc Substudy: Placebo | Total
Number analyzed (Participants) | 57 | 118 | 60 | 35 | 18 | 288
Age, Continuous [Mean (Full Range); unit: years] | 70.1 [46 to 83] | 70.4 [44 to 87] | 71.7 [39 to 85] | 69.7 [43 to 84] | 67.8 [54 to 81] | 69.9 [39 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 47 | 20 | 8 | 2 | 102
  Male | 32 | 71 | 40 | 27 | 16 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 5 | 0 | 0 | 12
  Not Hispanic or Latino | 48 | 100 | 48 | 29 | 15 | 240
  Unknown or Not Reported | 8 | 12 | 7 | 6 | 3 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 8 | 2 | 3 | 0 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 1 | 6
  White | 46 | 95 | 48 | 29 | 15 | 233
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 14 | 8 | 2 | 2 | 34

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Percentage of Participants Without Any Red Blood Cell (RBC) Transfusion During Any Consecutive 8-Weeks Period (All Participants)
Description: Percentage of participants without any RBC transfusion during any consecutive 8 weeks (56 days) starting from Study Day 1 until subsequent anti-cancer therapy if any were reported. Study Day 1 is defined as the day of the first dose for participants enrolled in Phase 2. The 95% confidence interval (CI) was calculated using Clopper-Pearson method. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 5 years in Phase 2
Population: Phase 2: All Treated Analysis Set included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Imetelstat Sodium
Number analyzed (Participants) | 57
percentage of participants | 36.8 [24.45 to 50.66]

2. Primary Outcome: Phase 2: Percentage of Participants Without Any RBC Transfusion During Any Consecutive 8-Weeks Period in Target Population
Description: as for outcome 1
Time Frame: Up to 5 years in Phase 2
Population: Phase 2: Target Population included participants without prior hypomethylating agent (HMA) or lenalidomide use and non del(5q) in karyotype at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Imetelstat Sodium
Number analyzed (Participants) | 38
percentage of participants | 42.1 [26.31 to 59.18]

3. Primary Outcome: Phase 3: Percentage of Participants Without Any RBC Transfusion During Any Consecutive 8-Weeks Period
Description: Percentage of participants without any RBC transfusion during any consecutive 8 weeks (56 days) starting from Study Day 1 until subsequent anti-cancer therapy if any were reported. Study Day 1 is defined as the day of the first dose for participants enrolled in Phase 2. The 95% CI was calculated using Clopper-Pearson method. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 3.7 years in Phase 3
Population: Phase 3: The ITT Analysis Set included all participants randomized into the Phase 3 study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 118 | 60
percentage of participants | 39.8 [30.93 to 49.25] | 15.0 [7.10 to 26.57]
Statistical Analysis 1: Comparison: Phase 3: Imetelstat Sodium vs Phase 3: Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The p-value was calculated based on Cochran-Mantel-Haenszel (CMH) controlling for prior RBC transfusion burden (≤6 versus[vs.]>6 units RBC) & international prognostic scoring system (IPSS) risk group (low vs. intermediate-1) applied to randomization; Percentage Difference = 24.8, 95% CI 2-sided [9.90 to 36.89] — The 95% CI was calculated based on the Wilson Score method

4. Secondary Outcome: Phase 2 and Phase 3: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Deaths
Description: TEAEs were defined as those events that 1) occurred after the first dose of study drug, through the treatment phase, and for 30 days following the last dose of study drug or until subsequent anti-cancer therapy if earlier; 2) any event that was considered study drug-related regardless of the start date of the event; or 3) any event that was presented at baseline but worsened in severity or was subsequently considered drug-related by the investigator. Serious TEAEs are any TEAEs that result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, is medically important. Any clinically significant vital sign measurements, clinical laboratory values, and electrocardiogram (ECG) findings were reported as TEAEs. TEAEs included both serious and non-serious TEAEs.
Time Frame: Adverse events: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3; Deaths: Up to 6.6 years in Phase 2 and up to 4 years in Phase 3
Population: Phase 2 and Phase 3: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Imetelstat Sodium (No Dose Escalation); Phase 3: Imetelstat Sodium: Imetelstat sodium administered IV, at a starting dose of 7.5 mg/kg, every 4 weeks (on a 28-day cycle) until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first.
- Phase 2: Imetelstat Sodium (Escalated to 9.4 mg/kg): Imetelstat sodium administered IV, at a starting dose of 7.5 mg/kg, every 4 weeks (on a 28-day cycle) with dose escalation to 9.4 mg/kg allowed before Protocol Amendment 2, until death, lost to follow up, withdrawal of consent, or study termination, whichever occurs first.
Arm/Group | Phase 2: Imetelstat Sodium (No Dose Escalation) | Phase 2: Imetelstat Sodium (Escalated to 9.4 mg/kg) | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 50 | 7 | 118 | 59
Participants
  Participants with AEs | 50 | 6 | 117 | 59
  Participants who died | 24 | 3 | 35 | 15

5. Secondary Outcome: Phase 2 and Phase 3: Percentage of Participants Without Any RBC Transfusion During Any Consecutive 24-Weeks Period
Description: Percentage of participants without any RBC transfusion during any consecutive 24 weeks (168 days) starting from Study Day 1 until subsequent anti-cancer therapy if any were reported. Study Day 1 is defined as the day of the first dose for participants enrolled in Phase 2 and the day of randomization for participants enrolled in Phase 3. The 95% CI was calculated using Clopper-Pearson method. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: Phase 2: All Treated Analysis Set included all participants who received at least one dose of study drug. Phase 3: ITT Analysis Set included all participants randomized into the Phase 3 study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 57 | 118 | 60
percentage of participants | 24.6 [14.13 to 37.76] | 28.0 [20.10 to 36.98] | 3.3 [0.41 to 11.53]
Statistical Analysis 1: Comparison: Phase 3: Imetelstat Sodium vs Phase 3: Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The p-value was calculated based on CMH controlling for prior RBC transfusion burden (≤6 vs. >6 units RBC) and IPSS risk group (low vs. intermediate-1) applied to randomization; Percentage Difference = 24.6, 95% CI 2-sided [12.64 to 34.18] — The 95% CI was calculated based on the Wilson Score method

6. Secondary Outcome: Phase 2 and Phase 3: Time to the 8-Weeks RBC Transfusion Independence (TI)
Description: Time to 8-week RBC TI was defined as the interval from Study Day 1 to the first day of the first 8-week RBC TI period.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: Phase 2: All Treated 8-week TI Responder Analysis Set included participants in the All Treated Analysis Set who achieved 8-week RBC TI.
  Phase 3: ITT 8-week TI Responder Analysis Set included all participants in the ITT Analysis Set who achieved 8-week RBC TI.
Measure: Median (Full Range); unit: weeks
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 21 | 47 | 9
weeks | 8.29 [0.1 to 100.6] | 9.29 [0.1 to 64.7] | 8.29 [0.1 to 46.9]

7. Secondary Outcome: Phase 2 and Phase 3: Time to the 24-Weeks RBC TI
Description: Time to 24-week RBC TI was defined as the interval from Study Day 1 to the first day of the first 24-weeks RBC TI period.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: Phase 2: All Treated 24-week TI Responder Analysis Set included participants in the All Treated Analysis Set who achieved 24-week RBC TI.
  Phase 3: ITT 24-week TI Responder Analysis Set included all participants in the ITT Analysis Set who achieved 24-week RBC TI.
Measure: Median (Full Range); unit: weeks
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 14 | 33 | 2
weeks | 8.79 [3.3 to 100.6] | 8.43 [2.1 to 37.6] | 3.79 [0.3 to 7.3]

8. Secondary Outcome: Phase 2 and Phase 3: Duration of RBC TI
Description: Duration of RBC TI was defined as the first day of the longest RBC TI period to the date of the first RBC transfusion after the TI period started. The 95% CI was based on Kaplan-Meier product limit estimates.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 21 | 47 | 9
weeks | 69.6 [17.00 to 92.43] | 51.6 [26.86 to 80.43] | 13.3 [8.00 to 24.86]
Statistical Analysis 1: Comparison: Phase 3: Imetelstat Sodium vs Phase 3: Placebo; Test type: Superiority; p < 0.001, Log Rank — The p-value (2-sided) was calculated using the stratified log-rank test for superiority of imetelstat sodium versus placebo in hazard ratio; Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.105 to 0.586] — Hazard ratio and 95% CI were calculated using the Cox proportional hazard model, stratified by prior RBC transfusion burden (≤ 6 vs. > 6 units RBC) and IPSS risk group (low vs. intermediate-1), with treatment as the only covariate

9. Secondary Outcome: Phase 2 and Phase 3: Percentage of Participants With Hematologic Improvement Including Erythroid Response (HI-E) as Per International Working Group (IWG) Response Criteria 2006
Description: As per IWG Response Criteria 2006: HI-E was defined as a hemoglobin (Hb) increase by greater than or equal to (≥)1.5 grams per deciliter (g/dL) relevant reduction of units of RBC transfusions by an absolute number of at least 4 RBC transfusion units/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks. Only RBC transfusions given for a Hb of less than or equal to (≤)9 g/dL pretreatment were counted in the RBC transfusion response evaluation. The 95% CI was calculated using Clopper-Pearson method. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 57 | 118 | 60
percentage of participants | 61.4 [47.57 to 74.00] | 63.6 [54.20 to 72.22] | 51.7 [38.39 to 64.77]
Statistical Analysis 1: Comparison: Phase 3: Imetelstat Sodium vs Phase 3: Placebo; Test type: Superiority; p = 0.112, Cochran-Mantel-Haenszel — The p-value was calculated based on CMH controlling for prior RBC transfusion burden (≤ 6 vs. > 6 units RBC) and IPSS risk group (low vs. intermediate-1) applied to randomization; Percentage Difference = 11.9, 95% CI 2-sided [-4.10 to 27.56] — 95% CI was calculated based on the Wilson Score Method

10. Secondary Outcome: Phase 2: Percentage of Participants With Complete Remission (CR), Partial Remission (PR), or Marrow Complete Remission (mCR) as Per International Working Group (IWG) Response Criteria 2006 as Assessed by the Investigator
Description: As per the IWG Response Criteria 2006, CR was defined as Bone marrow: ≤5% myeloblasts with normal maturation of all cell lines; Peripheral blood (PB): Hb ≥11 g/dL; platelets ≥100 x 10^9/dL; neutrophils ≥1.0 x 10^9/liter; blasts: 0%. PR was defined as Bone marrow: ≤5% myeloblasts and decrease by ≥50% over pretreatment; cellularity and morphology not relevant. mCR was defined as Bone marrow: ≤5% myeloblasts and decreased by ≥50% over pre-treatment PB. Percentages were rounded off to the nearest single decimal place. All participants in Phase 2 were evaluated by the Investigator for CR/PR/mCR regardless of bone marrow blasts at baseline.
Time Frame: Up to 5 years in Phase 2
Population: Phase 2: All Treated Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Imetelstat Sodium
Number analyzed (Participants) | 57
percentage of participants
  Percentage of participants with CR | 8.8
  Percentage of participants with PR | 0
  Percentage of participants with mCR | 12.3

11. Secondary Outcome: Phase 3: Percentage of Participants With CR, PR, or mCR as Per IWG Response Criteria 2006 as Assessed by the Independent Review Committee (IRC)
Description: As per the IWG Response Criteria 2006, CR was defined as Bone marrow: ≤5% myeloblasts with normal maturation of all cell lines; PB: Hb ≥11 g/dL; platelets ≥100 x 10^9/dL; neutrophils ≥1.0 x 10^9/liter; blasts: 0%. PR was defined as Bone marrow: ≤5% myeloblasts and decrease by ≥50% over pretreatment; cellularity and morphology not relevant. mCR was defined as Bone marrow: ≤5% myeloblasts and decreased by ≥50% over pre-treatment PB. CR, PR and mCR were assessed by IRC in Phase 3 and participants were required to fit at least one of the following criteria (participants with >5% baseline blasts per central pathology reviewer assessment; participants with CR, PR, mCR, or cytogenetic response as assessed by the investigator) and have at least one post-baseline assessment.
Time Frame: Up to 3.7 years in Phase 3
Population: Phase 3: ITT Analysis Set included all participants randomized into the Phase 3 study. Overall number of participants analyzed is the number of participants with >5% baseline bone marrow aspirate blasts per central pathology reviewer's assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 1 | 1
percentage of participants
  Percentage of participants with CR | 0 | 0
  Percentage of participants with PR | 0 | 0
  Percentage of participants with mCR | 0 | 0

12. Secondary Outcome: Phase 2 and Phase 3: Overall Survival (OS)
Description: OS was defined as the interval from Study Day 1 to death from any cause. Survival time of living participants was censored on the last date a participant is known to be alive or lost to follow-up. The Kaplan-Meier method was used to estimate overall survival.
Time Frame: Up to 6.6 years in Phase 2 and up to 4 years in Phase 3
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 57 | 118 | 60
months | 55.3 [39.16 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 40.4 [37.06 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | NA [32.16 to NA] — Median and upper limit of 95% CI were not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Phase 3: Imetelstat Sodium vs Phase 3: Placebo; Test type: Superiority; p = 0.949, Log Rank — P value (two-sided) for superiority of imetelstat sodium versus placebo in hazard ratio was calculated using stratified log-rank test; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.526 to 1.823] — Hazard ratio and 95% CI were calculated from the Cox proportional hazard model, stratified by prior RBC transfusion burden (≤6 vs. >6 units RBC) and IPSS risk group (low vs. intermediate-1), with treatment as the only covariate

13. Secondary Outcome: Phase 2 and Phase 3: Progression Free Survival (PFS)
Description: Progression free survival was defined as the time interval from study Day 1 to the first date of disease progression or death from any cause, whichever occurs first. Disease progression as per IWG criteria was defined as: at least one of the following: at least 50 % decrement from maximum response levels in granulocytes or platelets; reduction in hemoglobin by ≥1.5 g/dL; transfusion dependence.
Time Frame: Up to 6.6 years in Phase 2 and up to 4 years in Phase 3
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 57 | 118 | 60
months | 34.2 [25.10 to 39.29] | NA [29.24 to NA] — Median and upper limit of 95% CI were not estimable due to low number of participants with events. | NA [16.72 to NA] — Median and upper limit of 95% CI were not estimable due to low number of participants with events.

14. Secondary Outcome: Phase 2 and Phase 3: Time to Progression to Acute Myeloid Leukemia (AML)
Description: Time to progression to AML was defined as the interval from Study Day 1 to the date of AML diagnosis. Participants who did not progress to AML and were still alive at the cutoff date for the analysis or who withdrew from the study (withdrawal of consent or lost to follow-up), data was censored at the date of the last disease evaluation.
Time Frame: Up to 6.6 years in Phase 2 and up to 4 years in Phase 3
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 57 | 118 | 60
months | NA [41.36 to NA] — Median and upper limit of 95% CI were not estimable by Kaplan-Meir method due to low number of participants with events. | NA [NA to NA] — Median, lower limit and upper limit of 95% CI were not estimable by Kaplan-Meir method due to low number of participants with events. | NA [NA to NA] — Median, lower limit and upper limit of 95% CI were not estimable by Kaplan-Meir method due to low number of participants with events.

15. Secondary Outcome: Phase 2 and Phase 3: Amount of RBC Transfusions in the Best 8-week Interval
Description: Amount of RBC transfusions for 8-week interval was defined as the total number of RBC transfusion units in a given 8-week interval during study. The best 8-week interval is a post-baseline 8-week interval where the participant had the fewest post-Study Day 1 RBC transfusion units. A valid 8-week period must start before the date of last dose of study drug + 30 days or end of treatment (EOT) visit whichever occurs first and ends before the first transfusion in post-treatment follow-up or the first day of subsequent anti-cancer therapy whichever occurs first.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number of RBC transfusions units
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 57 | 118 | 60
number of RBC transfusions units | 3.0 (3.48) | 3.1 (3.62) | 3.4 (2.13)

16. Secondary Outcome: Phase 2 and Phase 3: Percent Change in RBC Transfusions Relative to Prior Transfusion Burden
Description: Relative percent change in RBC transfusions per 8-week = (amount of RBC transfusions per 8-week - prior RBC transfusion burden) / prior RBC transfusion burden multiplied by 100%. Prior RBC transfusion burden was defined as the maximum number of RBC units transfused over any consecutive 8 weeks prior to study entry.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 57 | 118 | 60
percent change | -62.5 (38.36) | -57.75 (50.220) | -51.01 (31.606)

17. Secondary Outcome: Phase 2 and Phase 3: Percentage of Participants Who Received Any Myeloid Growth Factors
Description: Percentage of participants who received any myeloid growth factors starting from Study Day 1 were reported. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 57 | 118 | 60
percentage of participants | 33 | 35.6 | 5.0

18. Secondary Outcome: Phase 2 and Phase 3: Duration of Myeloid Growth Factors Administration
Description: Duration of myeloid growth factor administered starting from Study Day 1 was reported.
Time Frame: Up to 5 years in Phase 2 and up to 3.7 years in Phase 3
Population: Phase 2: All Treated Analysis Set included all participants who received at least one dose of study drug.
  Phase 3: ITT Analysis Set included all participants randomized into the Phase 3 study. Overall number of participants analyzed is the number of participants who had at least 1 dose of myeloid growth factors in Phase 2 and Phase 3.
Measure: Median (Full Range); unit: weeks
Arm/Group | Phase 2: Imetelstat Sodium | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 19 | 42 | 3
weeks | 1.43 [0.1 to 118.0] | 0.71 [0.1 to 12.9] | 3.14 [0.1 to 10.0]

19. Secondary Outcome: Phase 2 and Phase 3: Maximum Observed Plasma Concentration (Cmax)
Description: As pre-specified in the statistical analysis plan (SAP), participants in the imetelstat sodium arm group of Phase 2 and Phase 3 were pooled for pharmacokinetic (PK) data collection and analyses in this outcome measure. PK parameters were determined by population PK model.
Time Frame: Pre-dose on Cycle 1 Day 1 and pre-dose on Day 1 of every 3 cycles from Cycle 4 up to Cycle 66 in Phase 2 and Cycle 34 in Phase 3 (each cycle length= 28 days)
Population: PK Parameter Analysis Set included all densely, and sparsely sampled participants who had received at least 1 dose of imetelstat sodium and who had sufficient data to calculate PK parameters for plasma imetelstat sodium. Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Groups:
- Phase 2 and Phase 3: Imetelstat Sodium: For Phase 2: Imetelstat sodium administered IV, at a starting dose of 7.5 mg/kg, every 4 weeks (on a 28-day cycle) until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first. Dose escalation to 9.4 mg/kg was allowed before Protocol Amendment 2.
  For Phase 3: Imetelstat sodium administered IV, at a starting dose of 7.5 mg/kg, every 4 weeks (on a 28-day cycle) until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first.
Arm/Group | Phase 2 and Phase 3: Imetelstat Sodium
Number analyzed (Participants) | 170
micrograms per milliliter (mcg/mL) | 89.5 (27.3)

20. Secondary Outcome: Phase 2 and Phase 3: Area Under the Drug Concentration-Plasma Time Curve From Time Zero to Time 28 Days (AUC0-28d)
Description: As pre-specified in the statistical analysis plan (SAP), participants in the imetelstat sodium arm group of Phase 2 and Phase 3 were pooled for PK data collection and analyses in this outcome measure. PK parameters were determined by population PK model.
Time Frame: Cycle 1 (Days 1 to 28) (Cycle duration= 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hour*micrograms per milliliter(h*mcg/mL)
Arm/Group | Phase 2 and Phase 3: Imetelstat Sodium
Number analyzed (Participants) | 170
hour*micrograms per milliliter(h*mcg/mL) | 559 (43.2)

21. Secondary Outcome: Phase 2 and Phase 3: Percentage of Participants With Anti-drug Antibodies (ADA) to Imetelstat Sodium
Description: As pre-specified in the SAP, participants in the imetelstat sodium arm group of Phase 2 and Phase 3 were pooled for immunogenicity data collection and analyses in this outcome measure. Percentages were rounded off to the nearest single decimal place.
Time Frame: as for outcome 19
Population: The Pharmacodynamic (PD) Analysis Set included all participants who had at least one quantifiable post-dose determination on biomarker, efficacy or safety parameters as defined in the related Pharmacodynamics analysis plan. Overall number of participants analysed signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 and Phase 3: Imetelstat Sodium
Number analyzed (Participants) | 166
percentage of participants | 16.9

22. Secondary Outcome: Phase 3: Medical Resource Utilization Assessed Based on Percentage of Participants With Outpatient Medical Encounters
Description: Outpatient medical encounters included various sites of care: a) emergency room (ER) visits, b) hospital outpatient visits, c) home care visit, d) visit to lab, e) visit to doctor's office, f) other visits. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 3.7 years in Phase 3
Population: Phase 3: ITT Analysis Set included all participants randomized into the Phase 3 study.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 118 | 60
percentage of participants | 39.0 | 38.3

23. Secondary Outcome: Phase 3: Medical Resource Utilization Assessed Based on Duration of Hospitalization
Description: Hospitalization included any medical encounter defined as hospice, hospital inpatient department, and intensive care unit (ICU). Hospitalizations without end dates were not counted in the calculation of length of stay. If any participant had multiple readmissions, duration was calculated as the sum of all hospital stays.
Time Frame: Up to 3.7 years in Phase 3
Population: Phase 3: ITT Analysis Set included all participants randomized into the Phase 3 study. Overall number of participants analyzed is the number of participants who were hospitalized.
Measure: Median (Full Range); unit: days
Arm/Group | Phase 3: Imetelstat Sodium | Phase 3: Placebo
Number analyzed (Participants) | 43 | 14
days | 8.0 [1 to 47] | 16.5 [1 to 75]

24. Secondary Outcome: QTc Substudy: Change From Baseline in QT Interval by Fridericia's Correction Method (ΔQTcF)
Description: Baseline was defined as the mean of the measured ECG intervals collected at 3 time points (-1 hour, -0.5 hour, and 0 hour) prior to treatment administration on Cycle 1 Day 1 (Cycle length= 28 days)
Time Frame: Baseline, Cycle 1, Day 1: 0.5, 1, 2, 4, 6, and 8 hours post-dose (cycle length= 28 days)
Population: The QTc substudy analysis set included all participants who participated in QTc substudy and received at least one dose of study drug, with measurements at baseline as well as on-treatment with at least 1 post-dose time point with a ΔQTcF value. By-time Point Analysis Set included each post-baseline time point that had a non-missing change-from-baseline observation. Number analysed is the number of participants with data available for analysis at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | QTc substudy: Imetelstat Sodium | QTc substudy: Placebo
Number analyzed (Participants) | 29 | 16
milliseconds (ms)
  Change at 0.5 hr post-dose | 4.2 (1.54) | 1.9 (2.09)
  Change at 1 hr post-dose | 5.4 (1.47) | 0.4 (2.00)
  Change at 2 hr post-dose | 5.5 (1.56) | 3.7 (2.12)
  Change at 4 hr post-dose | 1.8 (2.43) | 1.1 (3.28)
  Change at 6 hr post-dose: number analyzed (Participants) | 26 | 16
  Change at 6 hr post-dose | 1.7 (2.37) | -1.1 (3.12)
  Change at 8 hr post-dose: number analyzed (Participants) | 26 | 15
  Change at 8 hr post-dose | 2.3 (2.53) | -3.4 (3.36)

25. Other Pre Specified Outcome: Extension Phase: Number of Participants With AEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. AEs included clinically significant vital signs measurements, clinical laboratory values and electrocardiograms (ECGs) changes.
Time Frame: Up to approximately 3 years in the extension phase
Reporting Status: Not Posted, anticipated posting 2027-10

26. Other Pre Specified Outcome: Extension Phase: Overall Survival
Time Frame: Up to approximately 3 years in the extension phase
Reporting Status: Not Posted, anticipated posting 2027-10

27. Other Pre Specified Outcome: Extension Phase: Progression Free Survival (PFS) Survival
Description: Progression free survival will be assessed as the time interval from the end of the Phase 3 study until death, withdrawal of consent, study termination, or until a subject is lost to follow-up. As per IWG criteria disease progression is defined as: at least one of the following: at least 50 percent (%) decrement from maximum response levels in granulocytes or platelets; reduction in hemoglobin by greater than or equal to ≥1.5 g/dL; transfusion dependence.
Time Frame: Up to approximately 3 years in the extension phase
Reporting Status: Not Posted, anticipated posting 2027-10

ADVERSE EVENTS:
Time Frame: Adverse events: Up to 5 years in Phase 2; up to 3.7 years in Phase 3; up to 1.3 years in QTc substudy; All-cause mortality: Up to 6.6 years in Phase 2; up to 4 years in Phase 3; up to 1.6 years in QTc substudy
Description: Safety Analysis Set=all participants who received at least 1 dose of study drug. Safety data for Phase 2 arm has been reported separately for the participants without dose escalation and with dose escalation from 7.5 mg/kg to 9.4 mg/kg. QTc Substudy: Crossover arm includes AEs data after crossover from placebo to Imetelstat. Placebo arm included AE data for participants randomized to placebo prior to crossover.
Groups:
- QTc Substudy: Crossover Imetelstat Sodium: After a minimum of 2 treatment cycles (28-day cycle) if a participant had no significant change to pRBC transfusion burden or evidence of clinical benefit per Investigator, after discussion with the Sponsor the participant was crossed over from placebo to receive imetelstat sodium 7.5 mg/kg.
- QTc Substudy: Placebo: Imetelstat sodium matching placebo administered IV, every 4 weeks (on a 28-day cycle), until death, lost to follow-up, withdrawal of consent, or study termination whichever occurs first. If after a minimum of 2 treatment cycles a participant has no significant change to pRBC transfusion burden or evidence of clinical benefit per Investigator, after discussion with the Sponsor the participant, he/she may be permitted to start treatment with imetelstat sodium.
Arm/Group | Phase 2: Imetelstat Sodium (No Dose Escalation) | Phase 2: Imetelstat Sodium (Escalated to 9.4 mg/kg) | Phase 3: Imetelstat Sodium | Phase 3: Placebo | QTc Substudy: Imetelstat Sodium | QTc Substudy: Crossover Imetelstat Sodium | QTc Substudy: Placebo
All-Cause Mortality (participants affected / at risk) | 24/50 | 3/7 | 35/118 | 15/59 | 1/35 | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 26/50 | 1/7 | 41/118 | 13/59 | 8/35 | 3/14 | 0/18
Other Adverse Events (participants affected / at risk) | 50/50 | 6/7 | 117/118 | 58/59 | 33/35 | 12/14 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: Imetelstat Sodium (No Dose Escalation) (N=50) | Phase 2: Imetelstat Sodium (Escalated to 9.4 mg/kg) (N=7) | Phase 3: Imetelstat Sodium (N=118) | Phase 3: Placebo (N=59) | QTc Substudy: Imetelstat Sodium (N=35) | QTc Substudy: Crossover Imetelstat Sodium (N=14) | QTc Substudy: Placebo (N=18)
Pneumonia (Infections and infestations) | 2 | 0 | 3 | 1 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 2 | 3 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Corynebacterium infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermo-hypodermitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 1 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 0 | 1 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurodegenerative disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Kidney congestion (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: Imetelstat Sodium (No Dose Escalation) (N=50) | Phase 2: Imetelstat Sodium (Escalated to 9.4 mg/kg) (N=7) | Phase 3: Imetelstat Sodium (N=118) | Phase 3: Placebo (N=59) | QTc Substudy: Imetelstat Sodium (N=35) | QTc Substudy: Crossover Imetelstat Sodium (N=14) | QTc Substudy: Placebo (N=18)
Neutropenia (Blood and lymphatic system disorders) | 36 | 2 | 89 | 5 | 26 | 8 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 33 | 2 | 89 | 6 | 25 | 9 | 3
Anaemia (Blood and lymphatic system disorders) | 12 | 1 | 23 | 7 | 3 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 11 | 0 | 12 | 1 | 5 | 3 | 1
Pyrexia (General disorders) | 10 | 1 | 10 | 7 | 0 | 0 | 1
Oedema peripheral (General disorders) | 7 | 1 | 15 | 8 | 3 | 2 | 0
Fatigue (General disorders) | 5 | 2 | 9 | 4 | 5 | 2 | 1
Asthenia (General disorders) | 4 | 2 | 21 | 8 | 2 | 1 | 1
Influenza like illness (General disorders) | 2 | 2 | 0 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 0 | 0 | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 10 | 0 | 7 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 19 | 4 | 4 | 1 | 1
Chest pain (General disorders) | 2 | 0 | 2 | 5 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 0 | 11 | 5 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 0 | 1 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 10 | 1 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6 | 3 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 5 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 14 | 7 | 6 | 3 | 1
Constipation (Gastrointestinal disorders) | 8 | 0 | 10 | 7 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 0 | 9 | 3 | 2 | 3 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 8 | 2 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 2 | 4 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 7 | 3 | 13 | 4 | 6 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 2 | 11 | 4 | 3 | 3 | 1
Blood creatinine increased (Investigations) | 4 | 0 | 2 | 3 | 2 | 0 | 0
Headache (Nervous system disorders) | 11 | 2 | 15 | 3 | 3 | 1 | 1
Dizziness (Nervous system disorders) | 4 | 1 | 7 | 4 | 2 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0 | 2 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 1
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 0 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 2 | 3 | 3 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 11 | 6 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 9 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 5 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 3 | 1 | 7 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 3 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 0 | 0 | 0 | 4 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 6 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 7 | 1 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3 | 2 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serum ferritin increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Presbyacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melanoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consistent with Good Publication Practices and ICMJE guidelines, the sponsor shall have right to publish such primary (multicenter) data and information without approval from investigator. Investigator has right to publish study site-specific data after primary data published. If an investigator wishes to publish information from study, a copy of manuscript must be provided to sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT02598661/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT02598661/SAP_001.pdf